CLINICAL TRIAL: NCT07310160
Title: Development of a Digital Twin-Haptic Integrated Mixed Reality Simulation for Pressure Injury Management
Brief Title: Digital Twin-Haptic Integrated Mixed Reality Simulation
Acronym: DT-HIMRS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NEBAHAT BORA GÜNEŞ (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, NEBAHAT BORA GÜNEŞ, Assitant Professor, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 124S837; 124S834 (Other Grant/Funding Number: The Scientific and Technological Research Council of Türkiye (TÜBİTAK) under Grant No.1001-ID. 124S837)
Record Dates: First submitted 2025-12-04; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pressure Injury; Simulation Based Learning; Nursing
Keywords: haptic; mixed reality; digital twin
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Twin Haptic Integrated Simulation Group (Experimental): Participants in the digital twin-haptic integrated simulation group will receive training on pressure injury management using a virtual reality environment integrated with real-time digital twin and haptic feedback technologies. Nursing students who scored above 50 in the Fundamentals of Nursing course will be included. Those with communication barriers or balance disorders (e.g., vertigo) will be excluded. Participants who miss pre-, post-, or follow-up tests or fail to complete the intervention will be withdrawn. The intervention aims to enhance clinical reasoning, spatial awareness, and psychomotor skills through immersive, interactive simulation.
  Interventions: Device: Digital Twin-Haptic Integrated Simulation
- High-Fidelity Simulation Group (Active Comparator): Participants in the high-fidelity simulation group will engage in a pressure injury management training using the high-fidelity simulator (SimMan®) within the faculty's simulation laboratory. Nursing students who scored above 50 in the Fundamentals of Nursing course will be included. Those with communication barriers or balance disorders (e.g., vertigo) will be excluded. Participants who fail to attend pre-, post-, or follow-up tests or do not complete the simulation will be withdrawn. The intervention aims to improve clinical decision-making and psychomotor skills through realistic, hands-on simulation experience.
  Interventions: Behavioral: High-Fidelity Simulation

INTERVENTIONS:
Device: Digital Twin-Haptic Integrated Simulation — Participants perform pressure injury care procedures using a virtual reality simulation with a real-time digital twin and haptic feedback. Students wear VR headsets and interact with a digital model of the wound while performing physical actions such as wound assessment, cleansing, dressing, and patient repositioning. The digital twin mirrors each action to provide immediate visual and tactile feedback. This method allows students to practice clinical skills in a controlled environment, combining virtual and physical components. No brand-specific equipment names are used, and all activities follow established clinical guidelines.
  Arms: Digital Twin Haptic Integrated Simulation Group
Behavioral: High-Fidelity Simulation — Participants perform pressure injury care on a high-fidelity manikin in a simulation laboratory. The structured scenario includes wound assessment, cleansing, application of cream, dressing, and patient repositioning. The simulation replicates clinical procedures in a controlled setting, allowing students to practice and apply theoretical knowledge to standard nursing care. No brand-specific equipment names are used, and all activities follow established clinical guidelines.
  Arms: High-Fidelity Simulation Group

SUMMARY:
The responsibility for the management of pressure injuries belongs to nurses; the development of pressure injuries indicates that nursing care is not adequate. Pressure injury management should be addressed starting from undergraduate education in line with current guidelines. However, programs in which traditional education methods are used in pressure injury management are insufficient. Therefore, pressure injuries should be addressed with a structured simulation practice integrated with advanced technological methods. Any study using mixed reality in pressure injury management was not found in the literature. There is a study using augmented reality with a smartphone to measure wounds and a study examining the effectiveness of augmented reality in leg ulcer care. The use of mixed reality simulation in pressure injury management is one of the unique values of the project. Within the scope of the project, anchoring and monitoring physical objects in all application steps in pressure injury management and creating a digital twin is the most important original value of this project, which is that the student is immersed in the virtual reality environment in real-time and experiences all the processes physically-haptically. The digital twin-haptic integrated mixed reality simulation proposed in this project will contribute to the pressure injury literature and education by increasing the retention of information in memory and providing a realistic experience to the student, as it appeals to both visual, auditory, and tactile senses. The main aim of this project is to develop a digital twin-haptic integrated mixed reality simulation in pressure injury management and to compare the effect of the developed digital twin-haptic integrated mixed reality simulation and the high reality simulation in the institutional infrastructure on the students' knowledge level, skill performance, perceived learning level, satisfaction, and confidence level in learning. The project is planned as a randomized and comparative type and will last 24 months. A total of 130 second-year nursing undergraduate students will be stratified and randomized into the digital twin-haptic integrated mixed reality simulation and high-fidelity simulation groups based on their course grades and gender. Data will be collected using tests and scales. In terms of project management, the project has been handled in four phases with six work packages; in the first preparation phase, validity and reliability studies of the data collection tools, scenarios, and theoretical training module developed by the project team will be carried out, and participant randomization will be carried out. In the second phase, simulation laboratories will be prepared. In the third stage, the mixed-reality simulation software will be created and tested. In the last stage, pre-test application, training with the theoretical training module, simulation application, post-test, and follow-up will be carried out. Data will be analyzed using SPSS®23. All work to be carried out within the scope of the project is defined concretely and according to the workflow, and who/s will carry out each work is defined according to the field of expertise. All possible risks that may be encountered during the project have been foreseen, and measures for risk management have been prepared as Plan B. Within the scope of the project, importance was given to the use of the facilities, infrastructure, and equipment available in the institution. Within the scope of the project, the digital twin-haptic integrated mixed reality simulation will be developed entirely with national resources and registered. The mixed reality simulation software will be commercialized for educational purposes. In addition, with the use of the digital twin-haptic integrated mixed reality simulation program in the management of pressure injury, the quality of education in the field of health will increase, and the IT infrastructure of the training curricula will be supported, and a standard will be provided throughout the country, thus creating a sufficient and qualified workforce in this field. As a result of this qualified training, it is predicted that pressure injury rates will decrease and patient safety will increase in the long term. With the mixed reality simulation program, the leadership power of our country in the international arena, its potential, and recognition in the field of education and technology will be increased.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students enrolled in the Fundamentals of Nursing course.
* Students who achieved a score of 50 or higher in the Fundamentals of Nursing course.
* Students who voluntarily agree to participate in the study and provide informed consent.

Exclusion Criteria:

* Students with any communication barriers that may prevent participation or comprehension.
* Students with balance disorders (e.g., vertigo) or other medical conditions that could interfere with participation in the simulation.
* Students who fail to attend pre-test, post-test, or follow-up assessments.
* Students who do not participate in or complete the assigned simulation intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
Pressure Injury Management Skill Level | Pre-test, the day after intervention, 3-week follow-up
  Evaluates students' practical performances in pressure injury care, including wound assessment, cleansing, dressing, and patient repositioning with 6-item skill checklist based on NPIAP guidelines. Each item scored 0-1; total 0-6. Inter-rater reliability assessed via Kendall W coefficient.
Pressure Injury Management Knowledge Level | Pre-test, the day after intervention, 3-week follow-up
  Measures students' cognitive knowledge of pressure injury management with 20-item multiple-choice test. Each correct answer scores 1 point; total score ranges from 0 to 20. Test items were reviewed for content validity by experts and item analysis was performed to ensure reliability.

SECONDARY OUTCOMES:
Perceived Learning in Pressure Injury Care | Pre-test, the day after intervention, 3-week follow-up
  Measures students' self-reported learning in cognitive, affective, and psychomotor domains specifically related to pressure injury care. with a 9-item Rovai Perceived Learning Scale (cognitive, affective, psychomotor subscales) 7-point Likert scale; higher scores indicate higher perceived learning.
Satisfaction and Self-Confidence in Pressure Injury Training | Pre-test, the day after intervention, 3-week follow-up
  Assesses students' satisfaction with the pressure injury simulation (teaching methods, materials, facilitation) and their confidence in performing the learned skills, including wound care and clinical decision-making with 13-item NLN Student Satisfaction and Self-Confidence Scale. Items scored on 5-point Likert scale; higher scores indicate greater satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Özdemir, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaylor J, Hooper V, Wilson A, Burkert R, Lyda M, Fletcher K, Bowers E. Reliability Testing of Augmented Reality Glasses Technology: Establishing the Evidence Base for Telewound Care. J Wound Ostomy Continence Nurs. 2019 Nov/Dec;46(6):485-490. doi: 10.1097/WON.0000000000000585. PMID 31633610
- [Background] Hoenig, W., Milanes, C., Scaria, L., Phan, T., Bolas, M., & Ayanian, N. (2015, September). Mixed reality for robotics. In 2015 IEEE/RSJ International Conference on Intelligent Robots and Systems (IROS) (pp. 5382-5387). IEEE.
- [Background] Hauze SW, Hoyt HH, Frazee JP, Greiner PA, Marshall JM. Enhancing Nursing Education Through Affordable and Realistic Holographic Mixed Reality: The Virtual Standardized Patient for Clinical Simulation. Adv Exp Med Biol. 2019;1120:1-13. doi: 10.1007/978-3-030-06070-1_1. PMID 30919290
- [Background] Baratz G, Sridharan PS, Yong V, Tatsuoka C, Griswold MA, Wish-Baratz S. Comparing learning retention in medical students using mixed-reality to supplement dissection: a preliminary study. Int J Med Educ. 2022 Apr 29;13:107-114. doi: 10.5116/ijme.6250.0af8. PMID 35506483